CLINICAL TRIAL: NCT05203081
Title: Reliability and Validity of Urdu Version of National Institutes of Health Stroke Scale in Pakistani Stroke Population
Brief Title: Urdu Version of National Institutes of Health Stroke Scale: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00235
Record Dates: First submitted 2021-06-02; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: Stroke; Urdu version of National Institute of Health Stroke Scale; Reliability and Validity Study.; Glasgow Coma Scale; Modified Rankin Scale; Barthel Index
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study was to translate and culturally adapt NIHSS into Urdu language and to evaluate its reliability and validity in Pakistani stroke population. Also assess its correlation with Glasgow Coma Scale, Modified Rankin Scale and Barthel Index for severity and location of post-stroke impairment.

DETAILED DESCRIPTION:
As per preceding commendation, NIHSS has been translated into Urdu language from its English version and adapted culturally in Pakistan. Among stroke population, NIHSS-U has been administered in 225 patients recruited by convenience sampling technique under the pre-defined inclusion and exclusion criteria after signing consent forms. For testing inter-observer reliability and intra-observer reliability of NIHSS-U, GCS, mRS, and BI, questionnaires has been administered by two observers, on the same day, with a time interval of 2 hours between 1st and 2nd administration. As for the 3rd administration, it has been carried out after seven days by the first observer (re-testing), for intra-observer assessment. SPSS software version 24 has been used for the purpose of data entry and analysis. Internal consistency has been analyzed with Cronbach alpha value. Test-retest reliability has been assessed by using an intraclass correlation coefficient (ICC). The NIHSS-U has evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients or the ones next to them who gave informed consent.
* Age ranges from 34 to 97 years.
* Patients undertake particular stroke therapy including endovascular treatment intravenous thrombolysis.

Exclusion Criteria:

* Impaired strength of muscles because of cognitive and orthopedic diseases.
* Patients with severe hepatic, and/or renal diseases.
* Patients with impaired cognition and memory problems.
* Patients whose consent was not given by themselves, their caretakers.

Ages: 34 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We targeted the Pakistani stroke population with post-stroke impairments in our study.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | 1st day
  The National Institutes of Health Stroke Scale is a standardised evaluation tool for determining the neurological impairments that are most often encountered in acute stroke patients. It measures awareness, vision, visual fields, facial weakness, extremity motor performance, sensory deficiency, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect).
Glasgow Coma Scale | 1st day
  Glasgow Coma Scale is employed for patients suffering from head injury and has three components: eye opening, verbal response, and motor response. Score ranges from 3-15, lower score stands worse outcome
Modified Rankin Scale | 1st day
  Modified Rankin Scale is use to assess the degree of remaining disabilities while recovering from stroke. In mRS, 0-6 levels stands as; "0" for no symptom at all, "1" for no significant disability, "2" for slight disability, "3" for moderate disability, "4" for moderately severe disability, "5" for severe disability, and "6" for dead.
Barthel Index | 1st day
  Barthel Index is use to assess the level of independence and autonomy of stroke patient in performing ADLs. It is a list of 10 elementary ADLs: feeding, grooming, bathing, dressing, bowel and bladder care, toilet use, ambulation, transfers, and stair climbing. The activities are rated through time taken and assistance used by patient. Score ranges from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wisniewski A, Filipska K, Puchowska M, Piec K, Jaskolski F, Slusarz R. Validation of a Polish version of the National Institutes of Health Stroke Scale: Do moderate psychometric properties affect its clinical utility? PLoS One. 2021 Apr 2;16(4):e0249211. doi: 10.1371/journal.pone.0249211. eCollection 2021. PMID 33798218
- [Background] Sun TK, Chiu SC, Yeh SH, Chang KC. Assessing reliability and validity of the Chinese version of the stroke scale: scale development. Int J Nurs Stud. 2006 May;43(4):457-63. doi: 10.1016/j.ijnurstu.2005.07.004. Epub 2005 Sep 16. PMID 16146632
- [Background] Zhang S, Chang C, Zhang J, Song B, Fang H, Xu Y. Correlation analysis of sleep quality and youth ischemic stroke. Behav Neurol. 2014;2014:246841. doi: 10.1155/2014/246841. Epub 2014 Aug 5. PMID 25161340
- [Background] Banks JL, Marotta CA. Outcomes validity and reliability of the modified Rankin scale: implications for stroke clinical trials: a literature review and synthesis. Stroke. 2007 Mar;38(3):1091-6. doi: 10.1161/01.STR.0000258355.23810.c6. Epub 2007 Feb 1. PMID 17272767
- [Background] Kwon S, Hartzema AG, Duncan PW, Min-Lai S. Disability measures in stroke: relationship among the Barthel Index, the Functional Independence Measure, and the Modified Rankin Scale. Stroke. 2004 Apr;35(4):918-23. doi: 10.1161/01.STR.0000119385.56094.32. Epub 2004 Feb 19. PMID 14976324
- [Background] Nakao S, Takata S, Uemura H, Kashihara M, Osawa T, Komatsu K, Masuda Y, Okahisa T, Nishikawa K, Kondo S, Yamada M, Takahara R, Ogata Y, Nakamura Y, Nagahiro S, Kaji R, Yasui N. Relationship between Barthel Index scores during the acute phase of rehabilitation and subsequent ADL in stroke patients. J Med Invest. 2010 Feb;57(1-2):81-8. doi: 10.2152/jmi.57.81. PMID 20299746
- [Background] Ohura T, Hase K, Nakajima Y, Nakayama T. Validity and reliability of a performance evaluation tool based on the modified Barthel Index for stroke patients. BMC Med Res Methodol. 2017 Aug 25;17(1):131. doi: 10.1186/s12874-017-0409-2. PMID 28841846
- [Background] Hsueh IP, Lee MM, Hsieh CL. Psychometric characteristics of the Barthel activities of daily living index in stroke patients. J Formos Med Assoc. 2001 Aug;100(8):526-32. PMID 11678002
- [Background] Quinn TJ, Langhorne P, Stott DJ. Barthel index for stroke trials: development, properties, and application. Stroke. 2011 Apr;42(4):1146-51. doi: 10.1161/STROKEAHA.110.598540. Epub 2011 Mar 3. PMID 21372310
- [Background] Nik A, Sheikh Andalibi MS, Ehsaei MR, Zarifian A, Ghayoor Karimiani E, Bahadoorkhan G. The Efficacy of Glasgow Coma Scale (GCS) Score and Acute Physiology and Chronic Health Evaluation (APACHE) II for Predicting Hospital Mortality of ICU Patients with Acute Traumatic Brain Injury. Bull Emerg Trauma. 2018 Apr;6(2):141-145. doi: 10.29252/beat-060208. PMID 29719845